CLINICAL TRIAL: NCT01387841
Title: Comparison of Yoga Versus Relaxation on Chemotherapy Induced Nausea and Vomiting (CINV) Outcomes Following Chemotherapy
Brief Title: Effect of Yoga in Reducing Chemotherapy Induced Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bharath Charitable Cancer Hospital and Institute (Other)
Collaborators: Bangalore Institute of Oncology (Other); CENTRAL COUNCIL FOR RESEARCH IN YOGA AND NATUROPATHY (Unknown)
Responsible Party: Principal Investigator, Dr Raghavendra Rao M, Senior Scientist and Head CAM pROGRAM, Bharath Charitable Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Y010810
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer; Malignant Female Reproductive System Neoplasm; Lymphomas; Chemotherapy-induced Nausea and Vomiting
Keywords: yoga; chemotherapy; nausea; vomiting
MeSH Terms: conditions — Breast Neoplasms; Lymphoma; Vomiting; Nausea | interventions — Yoga

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Yoga group (Experimental): Yoga intervention with standard antiemetic care
  Interventions: Behavioral: yoga
- PMRT/Jacobsons Relaxation training (Active Comparator): 25 minutes of progressive muscle relaxation training will be given to this group with standard antiemetic care
  Interventions: Behavioral: Jacobsons PMRT group
- Standard antiemetic care (No Intervention): Standard antiemetic care only

INTERVENTIONS:
Behavioral: yoga — Postures,relaxation techniques
  Arms: Yoga group
Behavioral: Jacobsons PMRT group — jacobsons Progressive muscle relaxation training involving 16 muscle groups
  Other Names: PMRT
  Arms: PMRT/Jacobsons Relaxation training

SUMMARY:
* This randomized controlled three arm study compares the effects of a yoga intervention with jacobsons progressive muscle relaxation training and only standard of care in chemotherapy naive cancer patients.
* This study will also assess the neurophysiological correlates of nausea and vomiting and assess if effects of intervention on nausea and vomiting outcomes are mediated by changes in gastric motility (electrogastrogram) or stress arousal (cardiac autonomic function and sympathetic skin response) or self reported anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gynecologic malignancies (breast, ovary) and Lymphomas.
* Age between 30-70 years.
* Chemotherapy naïve.
* High school education.

Exclusion Criteria:

* Those with brain metastases
* Concurring medical condition likely to influence survival
* Uncontrolled diabetes and hypertension
* GI metastases, peritoneal fluid, uraemia
* Neurological disorders such as Parkinson's disease, myotonic dystrophy etc.
* GI obstruction and past H/o abdominal surgeries.
* Cognitive impairments.
* Regular participation in a behavioral intervention/yoga in the last six months

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Effect of yoga on chemotherapy induced nausea and vomiting | 4 months (prior to every cycle of chemotherapy,for 4 cycles)
  This study is to evaluate the effects of yoga intervention vs. Jacobsons progressive muscle relaxation vs. standard of care only on chemotherapy induced nausea and emesis (CINV) outcomes

SECONDARY OUTCOMES:
Quality of life after chemotherapy | 4 months
  Here we evaluate the effects of yoga intervention on secondary outcomes such as quality of life and anxiety states

CONTACTS AND LOCATIONS:
Overall Officials: RAGHAVENDRA RAO, PHD, Principal Investigator — HCG
Locations (1):
- Health Care Global, Bangalore, Karnataka, India